CLINICAL TRIAL: NCT05432531
Title: Efficiency of Baracetinib to Induce Remission of Active Lupus Nephritis
Brief Title: Efficiency of Use of Baracetinib in Treatment of Lupus Nephritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Associate Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Baracetinib
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Lupus Nephritis
MeSH Terms: conditions — Lupus Nephritis | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: patient and outcome assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Baracetinib (Experimental): oral tablet 4 mg baricitinib and placebo IV infusion/ month
  Interventions: Drug: Anti JAK1,2
- Cyclophosphamide (Active Comparator): IV cyclophosphamide 0.7mg/m2 every month and placebo tablet daily
  Interventions: Drug: Cyclophosphamid

INTERVENTIONS:
Drug: Anti JAK1,2 — Induction of remission of active lupus nephritis
  Other Names: Baritava
  Arms: Baracetinib
Drug: Cyclophosphamid — Induction of remission of active lupus nephritis
  Other Names: Indoxan
  Arms: Cyclophosphamide

SUMMARY:
Patients with systemic lupus erythematosus have substantial unmet medical need. Baricitinib is an oral selective Janus kinase (JAK)1 and JAK2 inhibitor that we hypothesised might have therapeutic benefit in patients with systemic lupus erythematosus and had a diagnosis of systemic lupus erythematosus, and had active renal disease as defined by Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K). Efficacy and safety analyses included all patients who received at least one dose of study drug.

DETAILED DESCRIPTION:
Patients with systemic lupus erythematosus have substantial unmet medical need. Baricitinib is an oral selective Janus kinase (JAK)1 and JAK2 inhibitor that we hypothesised might have therapeutic benefit in patients with systemic lupus erythematosus and had a diagnosis of systemic lupus erythematosus, and had active renal disease as defined by Systemic Lupus Erythematosus Disease Activity Index-2000 (SLEDAI-2K). Efficacy and safety analyses included all patients who received at least one dose of study drug.

The baricitinib 4 mg dose suggestive to significantly improved the signs and symptoms of active systemic lupus erythematosus in patients who were not adequately controlled despite standard of care therapy, with a safety profile consistent with previous studies of baricitinib. This study provides the idea for future trials of JAK1/2 inhibition with baricitinib as a new potential oral therapy for

ELIGIBILITY:
Inclusion Criteria:

* lupus nephritis

Exclusion Criteria:

* cardiac disease Thrombosis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Album in urine | 6 months
  24 h protein in urine

SECONDARY OUTCOMES:
complement 3 | 3 and 6 months
  serum level
anti double strand DNA | 3 and 6 months
  serum level
lupus activity index-2K | 3 and 6 months
  SLEDAI-2k

CONTACTS AND LOCATIONS:
Overall Officials: Manal M Hassanien, Md, Principal Investigator — Associate professor
Locations (1):
- Manal Hassanien, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No
After completing the study and published